CLINICAL TRIAL: NCT02302937
Title: A Prospective, Randomized, Controlled Trial to Compare Single Port Laparoscopic TEP Inguinal Hernia Repair Versus Standard Laparoscopic (3 Port) TEP Inguinal Hernia Mesh Repair
Brief Title: SIngle Port vs Standard TEP for Primary Inguinal Hernia Repair
Acronym: LESSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/00092; D/11/092 (Other: NUHS SIngapore)
Record Dates: First submitted 2013-12-05; First posted 2014-11-27 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2014-11

CONDITIONS: Primary Unilateral Inguinal Hernia
Keywords: Inguinal Hernia; Primary; laparoscopic surgery; single port surgery
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A: Standard TEP (Active Comparator): Group A will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm ).
  Interventions: Procedure: Group A will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm )
- Group B: LESS Port (Active Comparator): Group B will undergo laparoscopic TEP inguinal hernia repair with a single port (12 to 15 mm transumbilical).
  Interventions: Procedure: Group B will undergo laparoscopic TEP inguinal hernia repair with a single port

INTERVENTIONS:
Procedure: Group A will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm ) — laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm ).
  Arms: group A: Standard TEP
Procedure: Group B will undergo laparoscopic TEP inguinal hernia repair with a single port — Group B will undergo laparoscopic TEP inguinal hernia repair with a single port LESS (12 to 15 mm transumbilical).
  Arms: Group B: LESS Port

SUMMARY:
This study is carried out to determine if laparoscopic inguinal TEP repair of the hernia using a mesh carried out with only 1 port (hole) results in the reduction of post- operative pain and use of painkillers, shorter hospital stay and lesser complications than that carried out using conventional 3 ports.

DETAILED DESCRIPTION:
100 patients undergoing laparoscopic TEP ( Total extraperitoneal repair) inguinal hernia repair under general anaesthesia will be randomized into 2 groups by the closed envelope method. In case of difficulty in Single port TEP inguinal hernia repair, the procedure will be converted to conventional 3 port repair for patient safety.

2 groups of participants: Group A will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm ).

Group B will undergo laparoscopic TEP inguinal hernia repair with a single port (12 to 15 mm transumbilical).

Patient will be informed at consenting that 3 wound plasters will be applied to their abdomen regardless of whether they are in the single port or 3- ports group so that they would not know which group they have been randomized to. The blind will only be lifted after pain score and area of pain has been recorded before discharge.

ELIGIBILITY:
Inclusion Criteria:

Age: 21- 80 yrs

* Informed consent
* Diagnosis of Hernia
* ASA I and II
* BMI<25.

Exclusion Criteria:

Bleeding disorders

* Age below 21
* Strangulated Hernia
* BMI > 30
* Incarcerated and obstructed hernia
* Recurrent hernia
* Bilateral hernia
* Previous LSCS
* Previous lower abdominal surgery

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain score (Visual Analog Scale) at 24hours after surgery | 24 hours
  Assessment of post-operative pain according to the visual analog scale Pain score will be taken, and painkiller consumption will be recorded
Pain score (Visual Analog Scale) at 1 week after surgery | 1 week
  Assessment of pain according to the visual analog scale

SECONDARY OUTCOMES:
Recurrence of inguinal hernia | 1-3-6 months
  Finding of hernia again during examination after surgery
Post-operative complications | 1-3-6 months
  Examining for any seroma, hematoma and skin ecchymosis
Pain score (Visual Analog Scale) at 1-3-6 months after surgery | 1-3-6 months
  Assessment of pain according to the visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Piskun G, Rajpal S. Transumbilical laparoscopic cholecystectomy utilizes no incisions outside the umbilicus. J Laparoendosc Adv Surg Tech A. 1999 Aug;9(4):361-4. doi: 10.1089/lap.1999.9.361. PMID 10488834
- [Background] Goel R, Buhari SA, Foo J, Chung LK, Wen VL, Agarwal A, Lomanto D. Single-incision laparoscopic appendectomy: prospective case series at a single centre in Singapore. Surg Laparosc Endosc Percutan Tech. 2011 Oct;21(5):318-21. doi: 10.1097/SLE.0b013e3182311bd9. PMID 22002266
- [Background] Goo TT, Agarwal A, Goel R, Tan CT, Lomanto D, Cheah WK. Single-port access adrenalectomy: our initial experience. J Laparoendosc Adv Surg Tech A. 2011 Nov;21(9):815-9. doi: 10.1089/lap.2011.0179. Epub 2011 Sep 29. PMID 21958305
- [Result] Filipovic-Cugura J, Kirac I, Kulis T, Jankovic J, Bekavac-Beslin M. Single-incision laparoscopic surgery (SILS) for totally extraperitoneal (TEP) inguinal hernia repair: first case. Surg Endosc. 2009 Apr;23(4):920-1. doi: 10.1007/s00464-008-0318-x. Epub 2009 Jan 27. No abstract available. PMID 19172350
- [Derived] Chia DKA, Lomanto D, Wijerathne S. Patient-Reported Outcomes and Long-Term Results of a Randomized Controlled Trial Comparing Single-Port Versus Conventional Laparoscopic Inguinal Hernia Repair. World J Surg. 2020 Jul;44(7):2191-2198. doi: 10.1007/s00268-020-05443-z. PMID 32123978